CLINICAL TRIAL: NCT05235854
Title: Evaluation of the Performance of Six-month Wall Infiltration Under Ultrasound to Treat Stable Degenerative Meniscal Injuries. A Single-center, Randomized, Double-blind Study.
Brief Title: Six-month Performance of Meniscal Wall Infiltration Under Ultrasound to Treat Stable Degenerative Meniscal Injuries.
Acronym: ECHOGUIDE
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NIMAO/2021-1/PM-01
Record Dates: First submitted 2022-01-21; First posted 2022-02-11 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Osteoarthritis, Knee
Keywords: knee,; osteoarthritis,; meniscus,; Lysholm score,; corticoids; infiltration
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Intervention Model Description: Single-center, randomized, double-blind, controlled study comparing two management strategies.
Who Masked: Participant, Care Provider
Masking Description: The patient will not know whether he has been randomized to the meniscal wall infiltration group or the intra-articular filtration group. The investigator following up the patients after infiltration will not know whether his:her patient has had an intra-articular infiltration or a meniscal wall infiltration.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Meniscal wall infiltration group (Active Comparator): Administration of Diprostene: 1 ml syringe of Betamethasone 2 mg; injectable suspension in pre-filled syringe under ultrasound control.
  Interventions: Drug: Injection of corticosteroids (Diprostène®)
- Intra-articular infiltration group (Active Comparator): The procedure is identical in all respects to the experimental group, except that the ultrasound procedure is mimicked and the infiltration of dexamethasone 2 mg (Diprostene®) is performed intra-articularly.
  Administration Diprostene: 1 ml syringe of Betamethasone 2 mg; injectable suspension in pre-filled syringe.
  Interventions: Drug: Injection of corticosteroids (Diprostène®)

INTERVENTIONS:
Drug: Injection of corticosteroids (Diprostène®) — Diprostène® will be injected into the knee. This is a 1 ml syringe of Betamethasone 2 mg, suspension for injection in pre-filled syringe.

SUMMARY:
The main hypothesis of the study is that in situ infiltration of the meniscal lesion would provide patients with lasting and greater relief than intra-articular infiltration. A statistically significant difference would be if the Lysholm score of the meniscal wall group at 3 months is 9.5 points higher than that of the intra-articular infiltration group.

The aim is to evaluate the effectiveness of meniscal wall infiltration under ultrasound in the treatment of stable degenerative meniscal lesions versus intra-articular infiltration (Gold standard) at 3 months by Lysholm's algo-functional score.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a symptomatic meniscal lesion of a degenerative nature, isolated or associated with early osteoarthritis or chondropathy (Ahlbach stages 1 and 2).
* Indication for peri-meniscal infiltration under ultrasound control of the knee for a clinically stable degenerative meniscal lesion confirmed by MRI and radiography.
* Patient who has given free and informed consent.
* Patient who has signed the consent form.
* Patient affiliated or beneficiary of a health insurance plan.
* Adult patient (≥18 years of age).

Exclusion Criteria:

* No iconographic evidence of meniscal injury.
* Associated lesions of the central pivot of the knee.
* Knee pain of osteoarthritic origin strongly suggested by the clinic associated with an advanced radiological stage of osteoarthritis (Ahlbach stages 3 and 4).
* Presence of a skin lesion at the infiltration sites.
* Suspected soft tissue or joint infection.
* Patient participating in research involving human subjects defined as Category 1.
* Patient in an exclusion period as determined by another study.
* Patient under court protection, guardianship or trusteeship.
* Patient unable to give consent.
* Patient for whom it is impossible to give informed information.
* Pregnant, parturient or breastfeeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-05-12 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Lysholm score before infiltration (intra-articular group) | 15 days before infiltration
  The Lysholm score will be used to evaluate functionality 15 days before infiltration.The Lysholm Tegner score (Lysholm and Gillquist 1982) is a validated questionnaire for assessing knee functionality. The Lysholm score is rated from 0 to 100 (100 being the maximum functional score) and its repeatability is excellent (0.88 to 0.95). The scale has eight items: instability (/25), pain (/25), locking (/15), swelling (/10), stairs (/10), squatting (/5), limping (/5), use of a cane (/5). In 1985, Tegner added a scale of sports and occupational activity rated from 0 (occupational disability) to 10 (high level sport), hence the name Lysholm-Tegner score (Tegner and Lysholm 1985)
Lysholm score before infiltration (meniscal wall group) | 15 days before infiltration
  The Lysholm score will be used to evaluate functionality 15 days before infiltration.The Lysholm Tegner score (Lysholm and Gillquist 1982) is a validated questionnaire for assessing knee functionality. The Lysholm score is rated from 0 to 100 (100 being the maximum functional score) and its repeatability is excellent (0.88 to 0.95). The scale has eight items: instability (/25), pain (/25), locking (/15), swelling (/10), stairs (/10), squatting (/5), limping (/5), use of a cane (/5). In 1985, Tegner added a scale of sports and occupational activity rated from 0 (occupational disability) to 10 (high level sport), hence the name Lysholm-Tegner score (Tegner and Lysholm 1985)
Lysholm score after infiltration (intra-articular group) | 3 months after infiltration
  The Lysholm score will be used to evaluate functionality 3 months after infiltration.The Lysholm Tegner score (Lysholm and Gillquist 1982) is a validated questionnaire for assessing knee functionality. The Lysholm score is rated from 0 to 100 (100 being the maximum functional score) and its repeatability is excellent (0.88 to 0.95). The scale has eight items: instability (/25), pain (/25), locking (/15), swelling (/10), stairs (/10), squatting (/5), limping (/5), use of a cane (/5). In 1985, Tegner added a scale of sports and occupational activity rated from 0 (occupational disability) to 10 (high level sport), hence the name Lysholm-Tegner score (Tegner and Lysholm 1985)
Lysholm score after infiltration (meniscal wall group) | 3 months after infiltration
  The Lysholm score will be used to evaluate functionality 3 months after infiltration.The Lysholm Tegner score (Lysholm and Gillquist 1982) is a validated questionnaire for assessing knee functionality. The Lysholm score is rated from 0 to 100 (100 being the maximum functional score) and its repeatability is excellent (0.88 to 0.95). The scale has eight items: instability (/25), pain (/25), locking (/15), swelling (/10), stairs (/10), squatting (/5), limping (/5), use of a cane (/5). In 1985, Tegner added a scale of sports and occupational activity rated from 0 (occupational disability) to 10 (high level sport), hence the name Lysholm-Tegner score (Tegner and Lysholm 1985)

SECONDARY OUTCOMES:
Arthroscopy required within six months of infiltration: (intra-articular group) | 6 months after infiltration
  Yes/No and, if so, the date of the arthroscopy will be recorded.
Arthroscopy required within six months of infiltration: (meniscal wall group) | 6 months after infiltration
  Yes/No and, if so, the date of the arthroscopy will be recorded.
Pain evaluated by the patient (intra-articular group) | 15 days before infiltration
  Pain will be evaluated by the patient on a visual analog scale (0-10) once a week up to 3 months after infiltration.
Pain evaluated by the patient (intra-articular group) | 1 week after infiltration
  Pain will be evaluated by the patient on a visual analog scale (0-10) once a week up to 3 months after infiltration.
Pain evaluated by the patient (intra-articular group) | 2 weeks after infiltration
  Pain will be evaluated by the patient on a visual analog scale (0-10) once a week up to 3 months after infiltration.
Pain evaluated by the patient (intra-articular group) | 3 weeks after infiltration
  Pain will be evaluated by the patient on a visual analog scale (0-10) once a week up to 3 months after infiltration.
Pain evaluated by the patient (intra-articular group) | 4 weeks after infiltration
  Pain will be evaluated by the patient on a visual analog scale (0-10) once a week up to 3 months after infiltration.
Pain evaluated by the patient (intra-articular group) | 5 weeks after infiltration
  Pain will be evaluated by the patient on a visual analog scale (0-10) once a week up to 3 months after infiltration.
Pain evaluated by the patient (intra-articular group) | 6 weeks after infiltration
  Pain will be evaluated by the patient on a visual analog scale (0-10) once a week up to 3 months after infiltration.
Pain evaluated by the patient (intra-articular group) | 7 weeks after infiltration
  Pain will be evaluated by the patient on a visual analog scale (0-10) once a week up to 3 months after infiltration.
Pain evaluated by the patient (intra-articular group) | 8 weeks after infiltration
  Pain will be evaluated by the patient on a visual analog scale (0-10) once a week up to 3 months after infiltration.
Pain evaluated by the patient (intra-articular group) | 9 weeks after infiltration
  Pain will be evaluated by the patient on a visual analog scale (0-10) once a week up to 3 months after infiltration.
Pain evaluated by the patient (intra-articular group) | 10 weeks after infiltration
  Pain will be evaluated by the patient on a visual analog scale (0-10) once a week up to 3 months after infiltration.
Pain evaluated by the patient (intra-articular group) | 11 weeks after infiltration
  Pain will be evaluated by the patient on a visual analog scale (0-10) once a week up to 3 months after infiltration.
Pain evaluated by the patient (intra-articular group) | 12 weeks after infiltration
  Pain will be evaluated by the patient on a visual analog scale (0-10) once a week up to 3 months after infiltration.
Pain evaluated by the patient (meniscal wall group) | 15 days before infiltration
  Pain will be evaluated by the patient on a visual analog scale (0-10) once a week up to 3 months after infiltration.
Pain evaluated by the patient (meniscal wall group) | 1 week after infiltration
  Pain will be evaluated by the patient on a visual analog scale (0-10) once a week up to 3 months after infiltration.
Pain evaluated by the patient (meniscal wall group) | 2 weeks after infiltration
  Pain will be evaluated by the patient on a visual analog scale (0-10) once a week up to 3 months after infiltration.
Pain evaluated by the patient (meniscal wall group) | 3 weeks after infiltration
  Pain will be evaluated by the patient on a visual analog scale (0-10) once a week up to 3 months after infiltration.
Pain evaluated by the patient (meniscal wall group) | 4 weeks after infiltration
  Pain will be evaluated by the patient on a visual analog scale (0-10) once a week up to 3 months after infiltration.
Pain evaluated by the patient (meniscal wall group) | 5 weeks after infiltration
  Pain will be evaluated by the patient on a visual analog scale (0-10) once a week up to 3 months after infiltration.
Pain evaluated by the patient (meniscal wall group) | 6 weeks after infiltration
  Pain will be evaluated by the patient on a visual analog scale (0-10) once a week up to 3 months after infiltration.
Pain evaluated by the patient (meniscal wall group) | 7 weeks after infiltration
  Pain will be evaluated by the patient on a visual analog scale (0-10) once a week up to 3 months after infiltration.
Pain evaluated by the patient (meniscal wall group) | 8 weeks after infiltration
  Pain will be evaluated by the patient on a visual analog scale (0-10) once a week up to 3 months after infiltration.
Pain evaluated by the patient (meniscal wall group) | 9 weeks after infiltration
  Pain will be evaluated by the patient on a visual analog scale (0-10) once a week up to 3 months after infiltration.
Pain evaluated by the patient (meniscal wall group) | 10 weeks after infiltration
  Pain will be evaluated by the patient on a visual analog scale (0-10) once a week up to 3 months after infiltration.
Pain evaluated by the patient (meniscal wall group) | 11 weeks after infiltration
  Pain will be evaluated by the patient on a visual analog scale (0-10) once a week up to 3 months after infiltration.
Pain evaluated by the patient (meniscal wall group) | 12 weeks after infiltration
  Pain will be evaluated by the patient on a visual analog scale (0-10) once a week up to 3 months after infiltration.
Return to physical activity (intra-articular infiltration group) | Day 0 to Month 6
  The number of days taken for the patient to return to physical activity
Return to physical activity (meniscal wall infiltration group) | Day 0 to Month 6
  The number of days taken for the patient to return to physical activity
Adverse events in the intra-articular infiltration group | Day 0 to 3 months after infiltration
  Collection of all possible adverse events from D0 to M3. Qualitative
Adverse events in the meniscal wall infiltration group | Day 0 to 3 months after infiltration
  Collection of all possible adverse events from D0 to M3. Qualitative

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Nimes, Nîmes, France